CLINICAL TRIAL: NCT01222598
Title: Minirin Melt Tolerance With Nocturia in the Common Practice Conditions in Czech Republic
Brief Title: A Study of Minirin Melt in Patients With Nocturia
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE992026 CS38
Record Dates: First submitted 2010-10-05; First posted 2010-10-18 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a confirmation of safety profile for Minirin Melt in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from Nocturia

Exclusion Criteria:

* habitual or psychogenic polydipsia
* known or suspected cardiac insufficiency and other conditions requiring treatment with diuretics
* moderate and severe renal insufficiency
* know hyponatremia
* syndrome of inappropriate ADH secretion

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months

SECONDARY OUTCOMES:
Number of participants with nocturnal voiding | 12 months
Number of participants with adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (37):
- Czechia (37):
  - Private Ambulance, Blansko
  - Private Ambulance, Brno
  - Trauma Hospital in Brno, Brno
  - Urocentrum, Brno
  - Uromeda, s.r.o., Brno
  - Private Ambulance, Brno-Zábrdovice
  - Private Ambulance, Bystřice pod Hostýnem
  - Hospital Dečín, Děčín
  - University Hospital Hradec Králové, Hradec Králové
  - Hospital Jablonec nad Nisou, Jablonec nad Nisou
  - Hospital Jihlava, Jihlava
  - Hospital Kroměříž, Kroměříž
  - Polyclinic Kuřim, Kuřim
  - Private Ambulance, Moravský Krumlov
  - Hospital Nové Město na Moravě, Nové Město na Moravě
  - Hospital with Polyclinic Nový Jičín, Nový Jičín
  - Private Ambulance, Nový Jičín
  - University Hospital Olomouc, Olomouc
  - City Hospital Ostrava, Ostrava
  - Hospital Ostrava, Ostrava
  - Private Ambulance, Ostrava
  - Central Military Hospital, Prague
  - Medicon, s.r.o., Prague
  - Polyclinic Barandov, Prague
  - Private Ambulance, Prague
  - Railway Hospital, Prague
  - Thomayer´s Hospital, Prague
  - University Hospital Bulovka, Prague
  - Hospital Prostějov, Prostějov
  - Private Ambulance, Přerov
  - Hospital Šumperk, Šumperk
  - Private Ambulance, Třebíč
  - Hospital Uherské Hradiště, Uherské Hradiště
  - Hospital Ústí nad Orlicí, Inc, Ústí nad Orlicí
  - Hospital Valašské Meziříčí, Inc, Valašské Meziříčí
  - T. Bata Regional Hospital, Inc., Zlín
  - Hospital Znojmo, Znojmo